CLINICAL TRIAL: NCT04073589
Title: A Phase 1, Randomized, Open-label, Parallel-group Trial to Investigate the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Different Single Subcutaneous Dose Levels of Efgartigimod Co-administered With rHuPH20 in Healthy Adult Male Subjects
Brief Title: Efgartigimod Co-administered Subcutaneously With rHuPH20 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ARGX-113-1901; 2019-002102-40 (EudraCT Number)
Record Dates: First submitted 2019-08-16; First posted 2019-08-29 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Single SC injection of Dose A
  Interventions: Biological: ARGX-113 with rHuPH20
- Treatment B (Experimental): Single SC injection of Dose B
  Interventions: Biological: ARGX-113 with rHuPH20
- Treatment C (Experimental): Single SC injection of Dose C
  Interventions: Biological: ARGX-113 with rHuPH20
- Treatment D (Experimental): Single SC injection of Dose D
  Interventions: Biological: ARGX-113 with rHuPH20

INTERVENTIONS:
Biological: ARGX-113 with rHuPH20 — subcutaneous administration of efgartigimod with recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: efgartigimod with rHuPH20

SUMMARY:
The aim of this trial is to investigate the pharmacodynamic (PD), pharmacokinetic (PK), safety, tolerability, and immunogenicity of efgartigimod co-administered with rHuPH20, and to measure the time to inject the full dose of investigational medicinal product (IMP) of different dose levels of efgartigimod co-administered with a fixed concentration of rHuPH20 by the subcutaneous (SC) route of administration in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male, between 18 to 70 years of age
2. Subject is healthy
3. Subject has a body mass index (BMI) between 18 kg/m2 to 30 kg/m2
4. Subject is willing and able to understand the purpose and risks of the trial and provide signed and dated informed consent,
5. Others as defined in the protocol

Exclusion Criteria:

1. Previous participation in clinical trials with efgartigimod and/or any products with rHuPH20.
2. Known hypersensitivity to IMP ingredients or history of a severe allergic or anaphylactic reaction to any drug as determined by the investigator.
3. Known seropositivity or positive test at screening for an active viral infection with Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human immunodeficiency virus (HIV).
4. Known clinically relevant immunological disorders.
5. Known history or any symptom of clinically significant illness in the 6 months before IMP administration.
6. Others as defined in the protocol

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
IgG levels of four different subcutaneous dose levels | Up to 11 weeks, from study start until the end of the study

SECONDARY OUTCOMES:
Maximum serum concentrations (Cmax) of four different subcutaneous dose levels of efgartigimod co-administered with rHuPH20 | Up to 11 weeks, from study start until the end of the study
Time to reach maximum serum concentrations (Tmax) of four different subcutaneous dose levels of efgartigimod co-administered with rHuPH20 | Up to 11 weeks, from study start until the end of the study
Area Under The Curve (AUC) of four different subcutaneous dose levels of efgartigimod co-administered with rHuPH20 | Up to 11 weeks, from study start until the end of the study
Number of (serious) adverse events | Up to 11 weeks, from study start until the end of the study
Level of anti-drug antibodies | Up to 11 weeks, from study start until the end of the study
Time required to administer the different doses | Up to 11 weeks, from study start until the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guglietta, MD, Study Director — argenx
Locations (1):
- Investigator Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided